CLINICAL TRIAL: NCT06813066
Title: Simulating Psychotherapeutic Sessions With Generative Artificial Intelligence: A Proof-of-Concept Study of In Silico Psychotherapy Research
Brief Title: Simulating Psychotherapeutic Sessions With Generative Artificial Intelligence
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Trier University (Unknown); RWTH Aachen University (Other); University of Basel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 0000-00000; th24Meinlschmidt
Record Dates: First submitted 2025-02-03; First posted 2025-02-06 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Mental Disorder
Keywords: In silico Psychotherapy; Artificial intelligence (AI) applications; Motivational Interviewing
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Levels of Common Therapeutic Factors (Experimental): In this group, the patient-large language model (LLM) interacted with a therapist-LLM prompted to exhibit high levels of positive common factors.
  Interventions: Behavioral: High Levels of Common Therapeutic Factors
- Low Levels of Common Therapeutic Factors (Experimental): In this group, the patient-large language model (LLM) interacted with a therapist-LLM prompted to exhibit low levels of positive common factors.
  Interventions: Behavioral: Low Levels of Common Therapeutic Factors
- Transcripts of real intervention sessions (Other): This group consists of published transcripts of real intervention sessions, in which motivational interview techniques have been applied.
  Interventions: Behavioral: Standard motivational interviewing

INTERVENTIONS:
Behavioral: High Levels of Common Therapeutic Factors — The therapist large language model (LLM) is designed to show high levels of empathy, warmth, and genuineness. This setup aims to create a supportive and trusting therapeutic environment to improve patient engagement. High levels of these positive factors are linked to better psychotherapy outcomes and a stronger therapist-patient relationship.
  Arms: High Levels of Common Therapeutic Factors
Behavioral: Low Levels of Common Therapeutic Factors — The therapist LLM for this group is designed to show low levels of empathy, warmth, and genuineness. This setup aims to examine how a less supportive and empathetic therapist affects psychotherapy sessions. Lower levels of these positive behaviors can lead to reduced patient engagement and a weaker therapist-patient relationship, potentially hindering therapy outcomes.
  Arms: Low Levels of Common Therapeutic Factors
Behavioral: Standard motivational interviewing — Motivational interviewing techniques as applied during the sessions on which the transcripts are based.
  Arms: Transcripts of real intervention sessions

SUMMARY:
The study assesses the potential of using computational models, specifically large language models, to simulate psychotherapeutic sessions, aiming to improve therapy outcomes and advance therapist training through innovative technology.

DETAILED DESCRIPTION:
Health research has evolved significantly, increasingly incorporating computational models that improve our understanding and effectiveness of medical interventions. This shift from traditional to computational methods represents a major advancement in medical research, offering a more sustainable and innovative approach for conceptual advances and therapeutic discovery. In silico models, based on scientific simulation, use computational algorithms to mimic real-world systems or processes. This virtual environment allows researchers to explore phenomena impractical, unethical, dangerous, expensive, or impossible to study otherwise.

Psychotherapy is widely acknowledged as a primary treatment for a variety of mental health conditions, from depression and anxiety to personality disorders, offering significant pathways to recovery and improved quality of life. Yet current methods have shown limited effectiveness, prompting a need for innovative research approaches. In silico psychotherapy research leverages computational simulations, large language models (LLMs), and generative artificial intelligence to explore and refine psychotherapeutic interventions. By simulating human-like conversations, this approach provides insights into therapy dynamics and holds promise for revolutionizing therapist training and expanding treatment techniques.

This study aims to establish a proof-of-concept for simulating psychotherapeutic sessions using LLMs, focusing specifically on motivational interviewing. It involves the simulation of 512 psychotherapy sessions using LLMs as well as 8 real-world psychotherapy transcripts. By modeling human interactions, the study seeks to enhance healthcare delivery, therapist training, and personalized psychotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Simulation of psychotherapy sessions of conversations between an adult person presenting with a mental or behavioral health problem and a psychotherapist using large language models and 8 real-world transcripts

Exclusion Criteria:

* Simulation protocols with severe simulation errors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-04-26 (Estimated); Study Completion 2027-01-27 (Estimated)

PRIMARY OUTCOMES:
Simulation's Accuracy in generating Psychotherapeutic Dialogues | 12 months
  Assessment of the simulation's ability to accurately produce psychotherapeutic dialogues that adhere to the principles and techniques of motivational interviewing (MI), as determined by the average global scores of the Motivational Interviewing Treatment Integrity (MITI) code 4.2. The MITI code 4.2 includes various subscales, such as empathy and MI spirit, each scored on a scale from 1 to 5, with lower scores suggesting a need for improvement in MI delivery, while higher scores reflect stronger therapeutic skills and better patient outcomes.

SECONDARY OUTCOMES:
Number of Errors/Deviations | 12 months
  The number of errors or deviations from expected psychotherapeutic practices is counted, providing a quantitative measure of simulation quality. This measure also serves as exclusion criteria from any other assessment.
Metric of Verbal Content (Therapist) | 12 months
  Assessment of the text metrics of the therapist, based on the number of sentences, words, syllables, characters, and lexical diversity.
Metric of Verbal Content (Patient) | 12 months
  Assessment of the text metrics of the patient, based on the number of sentences, words, syllables, characters, and lexical diversity.
Turn-takings | 12 months
  Assessment of the turn-takings, based on the number of exchanges between the therapist and patient within a session, indicating the dynamic interaction flow.
Improvement of Patient | 12 months
  Improvement of the patient is evaluated using an an observer-rated, circularly framed version of the Importance and Confidence Rulers, measuring the simulated patient's psychotherapeutic progress on a circular scale from 0 to 10. Lower scores indicate lower perceived importance or confidence, while higher scores suggest greater perceived importance or confidence in making the change.
Credibility of Patient Behavior | 12 months
  The credibility of the patient's behavior is estimated using a 0 to 10 scale indicating how likely the evaluator found that the participants are real humans or simulations, offering insight into the perceived authenticity of the simulated interactions. The credibility of the 8 real-world transcripts served as a comparison baseline/benchmark for this evaluation. Lower scores indicate lower authenticity of the patient large-language model's (LLM's) simulated behavior, while higher scores suggest higher authenticity of the patient LLM's simulated behavior.
Credibility of Therapist Behavior | 12 months
  The credibility of the therapist's behavior is estimated using a 0 to 10 scale indicating how likely the evaluator found that the participants are real humans or simulations, offering insight into the perceived authenticity of the simulated interactions. The credibility of the 8 real-world transcripts served as a comparison baseline/benchmark for this evaluation. Lower scores indicate lower authenticity of the therapist large-language model's (LLM's) simulated behavior, while higher scores suggest higher authenticity of the therapist LLM's simulated behavior.
Manipulation Check | 12 months
  The implemented level of psychotherapeutic common factors by the therapist-LLM is approximated using the Therapist Empathy Scale (TES) as rough manipulation checks. The TES rates the therapist's ability to understand and share a patient's feelings on a scale from 1 to 7. Higher scores indicate greater empathy, reflecting a stronger connection and understanding of the patient's emotions, while lower scores suggest less empathy.
Manipulation Check | 12 months
  The implemented level of psychotherapeutic common factors by the therapist-LLM is approximated using the Working Alliance Inventory Short Observer form (WAI-S-O) as rough manipulation checks. The Working Alliance Inventory uses 12 items evaluating the perceived therapeutic alliance between the patient and the therapist on a scale of 1 to 7.

CONTACTS AND LOCATIONS:
Overall Officials: Gunther Meinlschmidt, Prof. Dr., Principal Investigator — University Hospital and University of Basel
Locations (1):
- University Hospital Basel, Basel, Switzerland